CLINICAL TRIAL: NCT07254182
Title: Effects of Ice-Pack Application on Hand Skin Temperature and Subjective Thermal Sensation and Comfort in Healthy Young Men: A Randomized, Parallel-Group Controlled Trial
Brief Title: Hand Cooling With Ice Packs in Healthy Young Men
Acronym: ICEHAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AWF-Poznan-HandIce-RCT-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Cold Exposure; Body Temperature Regulation; Thermal Comfort Perception
Keywords: Skin Temperature; Infrared Thermography (IRT); Thermal Sensation; Local Cooling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of outcomes assessors only. Thermographic image analysis and statistical analyses were performed by personnel not involved in data collection and blinded to group assignment; data were labeled by study ID without treatment identifiers. Participants and intervention administrators were unblinded due to perceptible cooling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice Pack (Localized Cryotherapy) (Experimental): Single 15-minute application of a reusable plastic ice pack (Mueller; Ø 22.86 cm, 946 mL). The pack was filled with 400 g of pre-portioned cylindrical ice and placed on the dorsal side of the dominant hand, ~1 cm proximal to the wrist-joint line, fully covering the fingers. Participants were supine with the hand slightly elevated; ambient conditions were controlled at ≈22.5 ± 1.0 °C and 55.3 ± 6.5% relative humidity (RH).Contact was maintained throughout the application; thermal sensation/comfort and pain were recorded during the 7th and 15th minutes.
  Interventions: Other: Ice Pack (Localized Cryotherapy)
- Thermoneutral Water Pack (Control) (Active Comparator): Identical 15-minute application using the same Mueller pack filled with thermoneutral water (within ±0.5 °C of limb skin temperature), mass-matched to 400 g. Placement, posture, and ambient conditions mirrored the experimental arm: pack on the dorsal side of the dominant hand, ~1 cm proximal to the wrist-joint line, fully covering the fingers; participants supine, hand slightly elevated; sensation/comfort and pain recorded at minutes 7 and 15.
  Interventions: Other: Thermoneutral Water Pack (Control)

INTERVENTIONS:
Other: Ice Pack (Localized Cryotherapy) — Single 15-minute application of a reusable plastic Mueller ice bag (Ø 22.86 cm, 946 mL). The bag was filled with 400 g pre-portioned cylindrical ice and placed on the dorsal side of the dominant hand, ~1 cm proximal to the wrist-joint line, fully covering the fingers. Participants were supine with the treated hand slightly elevated; ambient temperature and humidity were controlled (≈22.5 ± 1.0 °C; 55.3 ± 6.5% RH). Subjective thermal sensation/comfort (and pain) were recorded at minutes 7 and 15 during application. Arm: Experimental - Ice Pack
  Arms: Ice Pack (Localized Cryotherapy)
Other: Thermoneutral Water Pack (Control) — Identical 15-minute application using the same Mueller bag, filled with thermoneutral water (within ±0.5 °C of limb skin temperature), mass-matched to 400 g. Placement, posture, room conditions, and timing of subjective assessments (minutes 7 and 15) mirrored the experimental arm: bag on the dorsal side of the dominant hand, ~1 cm proximal to the wrist-joint line, fully covering the fingers; participants supine with the hand slightly elevated. Arm: Active Comparator - Thermoneutral Water Pack.
  Arms: Thermoneutral Water Pack (Control)

SUMMARY:
This randomized, parallel-group study looked at how a standard 15-minute ice pack applied to the back of the hand affects skin temperature and how cold and comfortable the hand feels, compared with a room-temperature water pack. Healthy young men were randomly assigned to one of the two groups during a single laboratory visit. Skin temperature was measured before, during, and after the application, and participants rated their thermal sensation (how cold/warm they felt) and overall comfort.

The main outcome was the change in hand skin temperature right after the 15-minute application. Additional outcomes included comfort and cold-feeling ratings and how quickly skin temperature returned toward baseline during recovery. This was a minimal-risk study; expected short-term effects included temporary cold, numbness, redness, or mild discomfort. No medicines or invasive procedures were used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers (university student population).
* Good general health with no history of neck or upper-quadrant pain.
* Able to provide written informed consent.
* Willing to comply with pre-visit restrictions on the study day (abstain from tobacco, coffee, alcohol; no hand ointments for 24 h; wash/degrease hands ≥1 h before testing; refrain from vigorous exercise/physical treatments for 24 h).

Exclusion Criteria:

* Diabetes
* Thyroid or other endocrine dysfunction
* Significant spinal pain
* Generalised neurological or rheumatological disorders
* Regular use of pain medications or psychotropic medications

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Minimum dorsal-hand skin temperature during rewarming (IV-X), by infrared thermography | From immediately after pack removal (0 minutes; time point IV) to 30 minutes after pack removal (time point X).
  Region-of-interest (ROI) mean skin temperature (Tsk; °C) on the dorsal hand measured with infrared thermography (IRT; FLIR SC640). The primary estimand is the between-group mean difference (Ice - Thermoneutral) in the nadir (minimum) across rewarming time points IV-X, with 95% confidence intervals (CI). Lower values indicate greater cooling.

SECONDARY OUTCOMES:
IRT-RT temperature offset at matched time points I-X | Baseline (after acclimatisation) and at 0, 5, 10, 15, 20, 25, and 30 minutes after ice-pack removal.
  Difference between infrared-thermography-derived skin temperature (TskIRT) and resistance temperature detector-derived skin temperature (TskRT), in degrees Celsius (°C), at each matched time point (I-X). IRT values represent ROI averages; resistance temperature (RT) values are point skin temperature readings from a RTD placed between the 3rd and 4th metacarpal bones. Positive values indicate that TskIRT is greater than TskRT. Between-group comparisons across time.
Change in Mechanical Detection Threshold (MDT) from baseline to immediately post (I → IV) | Baseline (after acclimatisation; time point I) and 0 minutes after ice-pack removal (time point IV).
  MDT (g) via Semmes-Weinstein monofilaments using an up-down procedure; analysed as IV - I. Higher values indicate reduced tactile sensitivity.
Change in Vibration Detection Threshold (VDT) from baseline to immediately post (I → IV) | Baseline (after acclimatisation; time point I) and 0 minutes after ice-pack removal (time point IV).
  VDT using a 64-Hz Rydel-Seiffer tuning fork (0-8/8 scale); analysed as IV - I. Higher values indicate reduced vibration sensitivity.
Thermal Sensation (TSS) during cooling and immediately post | Baseline (after acclimatisation; time point I), 7 minutes after ice-pack application (time point II), 15 minutes after ice-pack application (time point III), and 0 minutes after ice-pack removal (time point IV).
  9-point TSS (-4 very cold … +4 very hot) at I-IV; peak during cooling prespecified as the maximum at II or III. Between-group comparison of peak and trajectory.
Thermal Comfort (CS) during cooling and immediately post | Baseline (after acclimatisation; time point I), 7 minutes after ice-pack application (time point II), 15 minutes after ice-pack application (time point III), and 0 minutes after ice-pack removal (time point IV).
  5-point comfort scale (1 comfortable … 5 extremely uncomfortable) at I-IV; peak during cooling prespecified as the maximum at II or III.
Pain Intensity (Visual Analogue Scale; VAS) during cooling and immediately after ice-pack removal | Baseline (after acclimatisation; time point I), 7 minutes after ice-pack application (time point II), 15 minutes after ice-pack application (time point III), and 0 minutes after ice-pack removal (time point IV).
  0-100 mm visual analogue scale; peak during cooling prespecified as the maximum at II or III.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Straburzyńska-Lupa, MD, PhD, Study Chair — Department of Physical Therapy and Sports Recovery, Faculty of Health Sciences, Poznan University of Physical Education, 61-871 Poznań, Poland;; Pawel P Korman, PhD, Principal Investigator — Department of Physical Therapy and Sports Recovery, Faculty of Health Sciences, Poznan University of Physical Education, 61-871 Poznań, Poland;
Locations (1):
- Poznan University of Physical Education, Department of Physical Therapy and Sports Recovery, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available upon reasonable request for non-commercial research. Available IPD will include dorsal-hand skin temperature (IRT ROI means and RTD readings across time points I-X), thermal sensation, thermal comfort, pain VAS, MDT and VDT results, plus a data dictionary. Requests should be sent to [kontakt e-mail]. Proposals will be reviewed by the Principal Investigator; access requires a data use agreement and confirmation of ethics approval/waiver. Supporting materials (study protocol and SAP) and de-identified summary datasets are archived at Zenodo (DOI: 10.5281/zenodo.17255092).
Supporting Information: Study Protocol, SAP
Time Frame: From the date of article publication (or trial results posting) for 5 years.
Access Criteria: De-identified IPD (IRT skin temperature, RTD, thermal sensation/comfort, pain VAS, MDT, VDT, age [years], sex [male]) plus codebook available to qualified academic/non-profit researchers for non-commercial use. Request via email to [PI; pkorman@awf.poznan.pl] with a brief proposal and ethics approval; reviewed by the PI, response within 30 days. Access requires a Data Use Agreement (no re-ID, secure storage, no third-party sharing, use only as approved, cite the primary article/Zenodo, destroy/return within 5 years). Data provided as CSV via secure link after DUA; available from publication/results posting for up to 5 years; no fee.
URL: https://doi.org/10.5281/zenodo.17255092

REFERENCES:
- Available data/document: Individual Participant Data Set — https://zenodo.org/records/17255092
- Available data/document: Study Protocol — https://zenodo.org/records/17255092
- Available data/document: Statistical Analysis Plan — https://zenodo.org/records/17255092

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT07254182/Prot_SAP_000.pdf